CLINICAL TRIAL: NCT02203617
Title: Using Baby Books to Promote Maternal and Child Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Leonard Bickman, Professor, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD447749
Record Dates: First submitted 2014-07-18; First posted 2014-07-30 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Condition 1 - Educational Condition (Educational Book Group); Condition 2 - Non-educational Condition (Non-educational Book Group); Condition 3 - Control Condition (No-book Group)
Keywords: anticipatory guidance; baby books; safety

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- educational baby books (Experimental): books embedded with educational information (pediatric anticipatory guidance)
  Interventions: Behavioral: Educational Content/Pediatric Anticipatory Guidance; Behavioral: Book provision
- non-educational baby books (Active Comparator): baby books given with same illustrations but no educational information
  Interventions: Behavioral: Book provision
- no books (No Intervention): not given any baby books

INTERVENTIONS:
Behavioral: Educational Content/Pediatric Anticipatory Guidance — educational information from Bright Futures Guidelines for Health Supervision for birth to 18 months
  Arms: educational baby books
Behavioral: Book provision — Given free books prenatally and at 2, 4, 6, 9, 12, and 18 months postpartum
  Arms: educational baby books; non-educational baby books

SUMMARY:
The Baby Books Project tests whether embedding educational information into baby books can improve the health and wellbeing of first-time mothers and their young children.

DETAILED DESCRIPTION:
This study tests the efficacy of embedding educational information (i.e., pediatric anticipatory guidance) into baby books that first-time mothers read to their infants. This 3-group longitudinal study recruited first-time mothers in their third trimester of pregnancy, randomly assigned them to conditions, and followed them until the child was 18 months of age. One group received educational baby books, another group was given the same illustrated books with non-educational text, and the third group was not given any books. Thus, the effects of educational reading could be parsed from the effects of reading alone. The study aimed to test whether embedding pediatric anticipatory guidance in picture books is an effective method for increasing maternal knowledge of child development, parenting strategies, and safety practices, improving parenting beliefs and attitudes (e.g., parenting efficacy, importance of reading, use of corporal punishment), supporting optimal parenting practices (e.g., breastfeeding and nutrition, responsiveness, safety practices), improving maternal health (stress, depression), and supporting children's healthier development (injuries, illness, immunizations, and linguistic, social, and cognitive development).

Survey and observational data collection occurred in participants' homes during their third trimester of pregnancy and when their child was 2, 4, 6, 9, 12, and 18 months of age. Twelve phone call interviews were conducted between these home visits. When children were 18 months, a retrospective medical chart audit was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Women who are pregnant with first child and able to read in English at a first grade reading level

Exclusion Criteria:

* Women with other children, men, those not able to read in English at a first grade level

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2005-04; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of child development and parenting | Change from Baseline (pregnancy) to 18 months postpartum
  Measured with Opinions about Babies questionnaire
Change in Reading Practices | Change from 2 to 18 months postpartum
  Self-reported joint reading practices
Parenting Stress | Change from 2 to 18 months post-partum
  Measured with the Parenting Stress Index
Costs | Cumulative costs over study duration
  Maternal costs due to their own and their child's illness/injury, use of substances, and purchase of food was measured with the Incurred Cost Questionnaire.

SECONDARY OUTCOMES:
Safety Practices | 2, 4, 6, 9, 12, and 18 months postpartum
  Measured with the Home Safety Assessment, an observational and self-report measure of safety practices in the home, car, and outside
Attitudes about Corporal punishment | 2, 6, 12 and 18 months postpartum
  Adolescent-Adult Parenting Inventory
Maternal Depressive Symptoms | Change from baseline (pregnancy) to 18 months postpartum
  Depressive symptoms were measured with the Center for Epidemiologic Studies Depression Scale.
Beliefs about the Importance of Reading to Children | Change from baseline (prenatal) to 18 months postpartum
  Maternal beliefs about the importance of reading was measured with the Modified Parent Reading Belief Inventory
Injuries and illnesses | 16 months (from 2 to 18 months postpartum)
  Child illnesses injuries were measured with the Incurred Cost Questionnaire and through a retrospective medical chart audit.
Quality of Parent-Child Interaction | Change from 2 to 18 months postpartum
  Video recording and in-vivo coding of mother-child dyads during play and reading.
Home environment and parenting | Change from 2 to 18 months postpartum
  measured with the Home Observation for Measurement of Environment (HOME).
Receptive and Expressive language | Change from 6 to 18 months postpartum
  Measured with the Preschool Language Scale - Fourth Edition (PLS4).
Cognitive and neurological development screening | 4, 6, 9 months postpartum
  Measured with the Bayley Infant Neurodevelopmental Screener (BINS)
Infant nutrition | 2, 4, 6, 9, 12, and 18 months postpartum
  Infant Nutrition Interview measured the introduction of news foods, types of foods, and serving portions at each time point.
Breastfeeding intentions and practices | prenatal and postnatal every visit until no longer breastfeeding
  measured with the Breastfeeding Intentions and Practices Scale
Pregnancy uplifts and Hassles | Baselines (pregnancy)
  measured with the Pregnancy Experience Scale
Parenting Satisfaction | Change from 2 to 18 months postpartum
  measured with the Parenting Satisfaction Scale
Parenting Self-Efficacy | Change from 2 to 18 months postpartum
  Measured with the Maternal Self-Efficacy Scale
Reading self-efficacy | Change from 2 to 18 months postpartum
  measured with the Reading Self-Efficacy Scale
Cognitive Development | 12 and 18 months postpartum
  measured with Exploratory Play Task
Immunizations, medical visits, and growth status | 18 months postpartum
  measured through a retrospective medical chart audit.

OTHER OUTCOMES:
Community Conditions | 4 months postpartum and following a move to a new residence
  measured with the observational Community Conditions Checklist and self-report Community Conditions Interview

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M Reich, PhD, Study Director — University of California, Irvine; Leonard Bickman, PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Khalessi A, Reich SM. A Month of Breastfeeding Associated with Greater Adherence to Pediatric Nutrition Guidelines. J Reprod Infant Psychol. 2013 Jul 1;31(3):299-308. doi: 10.1080/02646838.2013.784898. PMID 24062596
- [Result] Reich SM, Penner EK, Duncan GJ, Auger A. Using baby books to change new mothers' attitudes about corporal punishment. Child Abuse Negl. 2012 Feb;36(2):108-17. doi: 10.1016/j.chiabu.2011.09.017. Epub 2012 Mar 3. PMID 22391417
- [Result] Reich SM, Penner EK, Duncan GJ. Using baby books to increase new mothers' safety practices. Acad Pediatr. 2011 Jan-Feb;11(1):34-43. doi: 10.1016/j.acap.2010.12.006. PMID 21272822
- [Result] Reich SM, Bickman L, Saville BR, Alvarez J. The effectiveness of baby books for providing pediatric anticipatory guidance to new mothers. Pediatrics. 2010 May;125(5):997-1002. doi: 10.1542/peds.2009-2728. Epub 2010 Apr 12. PMID 20385630